CLINICAL TRIAL: NCT06595615
Title: Health App Data Collection Study
Status: Not yet recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Huntsville Hospital Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 10470
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cardiovascular implantable electronic devices — Standard of care patients indicated for the devices

SUMMARY:
Utilization of additional wearable data to improve clinical outcome

DETAILED DESCRIPTION:
In addition to information available from cardiac implantable medical devices, health related data available from commercially approved wearables and devices such as Apple watch, blood pressure monitor and scales could be used to improve predictive analytics of impending clinical events. This study is to merge implantable medical device data with wearable data to evaluate the added benefit of extra data.

ELIGIBILITY:
Inclusion Criteria:

* Patients are willing to be compliant with daily measurements required 18 years of age or older
* Patients who have been implanted with ABT CRT-D devices connected to Merlin.net
* Patients who had at least one HF clinical event during past 12 calendar months
* Must provide written informed consent prior to the commencement of this clinical feasibility study
* Patients are willing to be compliant with daily measurements required

Exclusion Criteria:

* Pregnant and/or lactating mothers will be excluded from the study or have a plan to be pregnant in the next 12 months
* Patients with a life expectancy less than the duration of the study, as per clinician's discretion.
* Patients who will not be able to complete the daily survey questions due to inability to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for cardiac implantable medical devices
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acquisition of additional health data using patient App | 12 months
  Health data acquisition via an app from multiple wearables and externals.

IPD SHARING:
Plan to Share IPD: No